CLINICAL TRIAL: NCT05058547
Title: An Evidence-based Digital Support for One Year to Facilitate a Sustainable Return to Work for Persons With Chronic Musculoskeletal Pain and Their Employers: Study Protocol for a Registry-based Multicentre Randomized Controlled Trial.
Brief Title: A Digital Support to Facilitate Sustainable Return to Work for Persons With Chronic Pain and Their Employers
Acronym: SWEPPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Linkoeping University (Other Government)
Collaborators: Swedish Council for Working Life and Social Research (Other)
Responsible Party: Principal Investigator, Mathilda Björk, Deputy Head of Department, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr 2019-01264
Record Dates: First submitted 2021-09-24; First posted 2021-09-27 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Chronic Pain
Keywords: collaboration support; eHealth; employer support; smartphone application; return to work; self-management
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SWEPPE (Experimental): Participants will receive the smartphone application SWEPPE.
  Interventions: Device: SWEPPE
- Control (No Intervention): Participants randomized to the control group will not receive any active intervention for return to work after completing an Interdisciplinary Pain Rehabilitation Program .

INTERVENTIONS:
Device: SWEPPE — In the smartphone application SWEPPE the individual can create an action plan, perform daily registrations of health aspects, self-monitoring of health aspects and goals, have access to a library with evidence-based facts and a coach, and possibility to share information with the employer.
  Arms: SWEPPE

SUMMARY:
Chronic musculoskeletal pain (CMSP) severely affects the individual's quality of life, functioning and ability to work, and comes with significant societal costs for sick leave and loss of productivity. After completing an Interdisciplinary Pain Rehabilitation Program (IPRP), patients with CMSP experience a gap in the return to work (RTW) process when the responsibility for RTW is taken over by the employer. To fill this gap, we aim to evaluate the clinical effectiveness of a digital support (SWEPPE) for promoting a sustainable RTW for persons with CMSP and to facilitate the employers' supportive role and responsibilities in the process. Our hypothesis is that using SWEPPE will decrease the need for sick-leave.

SWEPPE is a smartphone application where the individual can create an action plan, perform daily registrations of health aspects, self-monitoring of health aspects and goals, have access to a library with evidence-based facts and a coach, and the possibility to share information with the employer.The employer access SWEPPE via a web application.

In this trial, we will recruit patients with CMSP aged 18-65 years who have completed IPRP, and who need support during RTW or continued support at the work placement for creating a sustainable work situation. The participants will be randomly assigned to either receive SWEPPE or to the control group. The intervention group will use SWEPPE during twelve months and the control group will not receive any active intervention for RTW which is standard clinical practice. Participants will be recruited from specialist and primary care level units connected to the Swedish National Quality Registry for Pain Rehabilitation (SQRP) and providing IPRP for patients with CMSP.

All participants will fill in questionnaires when they have completed the rehabilitation program and before the intervention starts. Study ending assessment will be performed after twelve months.

The clinical effectiveness of SWEPPE will be assessed by number of days with sickness cash benefit. Several dimensions of sick-leave will be assessed according to the Swedish Social Insurance Agency's (SSIA) proposal of outcome measures of RTW. Other outcomes and explanatory variables including important domains affected by CMSP such as health-related quality of life, functioning and work ability will be collected. A sample size calculation indicates the need for recruiting 360 participants (n=180 for each group).

ELIGIBILITY:
Inclusion Criteria:

Patients entering the trial must have completed IPRP. The principal inclusion criteria for IPRP in Sweden are:

* persistent or intermittent pain lasting ≥3 months
* pain affecting daily activities to a large extent,
* completed systematic assessment and non-pharmacological optimization is completed,
* screening for psychosocial risk factors and differential diagnosis completed

In addition the following criteria will be applied:

* Completed participation in an Interdisciplinary Pain Rehabilitation Program (IPRP) at any of the participating units.
* Having an employment to return to after IPRP or having returned to work but need continued support for creating a sustainable work situation after IPRP.

Exclusion criteria:

* Completed IPRP but are unemployed or unable to return to work.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Sick leave | 12 months follow up after IPRP
  Number of gross and net days with sickness cash benefit

SECONDARY OUTCOMES:
Return to work | 12 months follow up after IPRP
  Return to work (partially or full time) every month
Sick-leave spells per months | 12 months follow up after IPRP
  Number of sick-leave spells (per month)
Return to work group level | 12 months follow up after IPRP
  Proportions of a group who returns to full- or part-time work (per month)
Working days before new sick leave | 12 months follow up after IPRP
  Number of days in work before new sick leave during study period
Proportion back to work | 12 months follow up after IPRP
  Proportion of a group back to work >28 days (full- or part time) before a new sick-leave spell occurs
Total sick-leave spells | 12 months follow up after IPRP
  Number of sick-leave spells during study period
Length of total sick leave | 12 months follow up after IPRP
  Length of total sick leave during study period
Pain intensity last 7 days | Baseline and 12 months
  Numeric rating scale
Consequences of pain on daily life | Baseline and 12 months
  Multidimensional Pain Inventory Swedish version
Overall emotional distress | Baseline and 12 months
  Hospital Anxiety and Depression Scale Swedish version
Physical and mental health | Baseline and 12 months
  RAND-36 Swedish version
Goal fulfilment and satisfaction during the study period | Baseline and 12 months
  Self-reported data
Self-reported physical work environment | Baseline and 12 months
  Questionnaire based on the Swedish Work Environment Authority ergonomics checklist

OTHER OUTCOMES:
Self-reported fatigue the last 7 days | Baseline and 12 months
  Numeric rating scale
Self-reported level of sleepiness | Baseline and 12 months
  Karolinska Sleepiness Scale Swedish version
Self-reported level of sleep disturbance | Baseline and 12 months
  Insomnia Severity Index Swedish version
Self-reported fear of movement | Baseline and 12 months
  Tampa Scale for Kinesiophobia Swedish version
Self-reported physical activity | Baseline and 12 months
  the National Board of Health and Welfare's three questions on physical activity, exercise, and sedentary behavior.
Pain catastrophizing | Baseline and 12 months
  Pain Catastrophizing scale Swedish version
Perceived work ability | Baseline and 12 months
  Work Ability Index Swedish version
Self-reported demands, control, and support at the workplace | Baseline and 12 months
  Demand Control Support Questionnaire Swedish version
Perceived life Satisfaction | Baseline and 12 months
  Life satisfaction Scale Swedish version
Self-reported work situation during the study period | Baseline and 12 months
  Barriers for return to work, strategies to handle barriers and need of support from the employer
Self-reported workload an average day | Baseline and 12 months
  Number of hours per day for paid work and unpaid household work

CONTACTS AND LOCATIONS:
Overall Officials: Mathilda Björk, PhD, Principal Investigator — Linkoeping University
Locations (5):
- Sweden (5):
  - Danderyd hospital, Danderyd
  - Smärtcentrum, Karlstad
  - County council of Ostergotland, Linköping
  - Smärtcentrum, Lund
  - Spine Center, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harker J, Reid KJ, Bekkering GE, Kellen E, Bala MM, Riemsma R, Worthy G, Misso K, Kleijnen J. Epidemiology of chronic pain in denmark and sweden. Pain Res Treat. 2012;2012:371248. doi: 10.1155/2012/371248. Epub 2012 May 23. PMID 22693667
- [Background] Reid KJ, Harker J, Bala MM, Truyers C, Kellen E, Bekkering GE, Kleijnen J. Epidemiology of chronic non-cancer pain in Europe: narrative review of prevalence, pain treatments and pain impact. Curr Med Res Opin. 2011 Feb;27(2):449-62. doi: 10.1185/03007995.2010.545813. Epub 2011 Jan 3. PMID 21194394
- [Background] Perez C, Margarit C, Sanchez-Magro I, de Antonio A, Villoria J. Chronic Pain Features Relate to Quality of Life More than Physiopathology: A Cross-Sectional Evaluation in Pain Clinics. Pain Pract. 2017 Sep;17(7):866-878. doi: 10.1111/papr.12533. Epub 2017 Feb 25. PMID 27782366
- [Background] Gerdle B, Bjork J, Henriksson C, Bengtsson A. Prevalence of current and chronic pain and their influences upon work and healthcare-seeking: a population study. J Rheumatol. 2004 Jul;31(7):1399-406. PMID 15229963
- [Background] Caceres-Matos R, Gil-Garcia E, Barrientos-Trigo S, Porcel-Galvez AM, Cabrera-Leon A. Consequences of Chronic Non-Cancer Pain in adulthood. Scoping Review. Rev Saude Publica. 2020 Apr 17;54:39. doi: 10.11606/s1518-8787.2020054001675. eCollection 2020. PMID 32321056
- [Background] Asmundson GJ, Katz J. Understanding the co-occurrence of anxiety disorders and chronic pain: state-of-the-art. Depress Anxiety. 2009;26(10):888-901. doi: 10.1002/da.20600. PMID 19691031
- [Background] Shupler MS, Kramer JK, Cragg JJ, Jutzeler CR, Whitehurst DGT. Pan-Canadian Estimates of Chronic Pain Prevalence From 2000 to 2014: A Repeated Cross-Sectional Survey Analysis. J Pain. 2019 May;20(5):557-565. doi: 10.1016/j.jpain.2018.10.010. Epub 2018 Nov 29. PMID 30503860
- [Background] Svanholm F, Liedberg GM, Lofgren M, Bjork M. Factors of importance for return to work, experienced by patients with chronic pain that have completed a multimodal rehabilitation program - a focus group study. Disabil Rehabil. 2022 Mar;44(5):736-744. doi: 10.1080/09638288.2020.1780479. Epub 2020 Jun 25. PMID 32580604
- [Background] Toye F, Seers K, Allcock N, Briggs M, Carr E, Barker K. A synthesis of qualitative research exploring the barriers to staying in work with chronic musculoskeletal pain. Disabil Rehabil. 2016;38(6):566-72. doi: 10.3109/09638288.2015.1049377. PMID 26017361
- [Background] Liedberg GM, Bjork M, Dragioti E, Turesson C. Qualitative Evidence from Studies of Interventions Aimed at Return to Work and Staying at Work for Persons with Chronic Musculoskeletal Pain. J Clin Med. 2021 Mar 17;10(6):1247. doi: 10.3390/jcm10061247. PMID 33802906
- [Background] Saunders SL, Nedelec B. What work means to people with work disability: a scoping review. J Occup Rehabil. 2014 Mar;24(1):100-10. doi: 10.1007/s10926-013-9436-y. PMID 23519737
- [Background] Grant M, O-Beirne-Elliman J, Froud R, Underwood M, Seers K. The work of return to work. Challenges of returning to work when you have chronic pain: a meta-ethnography. BMJ Open. 2019 Jun 20;9(6):e025743. doi: 10.1136/bmjopen-2018-025743. PMID 31227529
- [Background] Magalhães L, Chan C, Chapman A, Majed L, Samigullina R, Trninic D, et al. Successful return to work of individuals with chronic pain according to health care providers: a meta-synthesis. Cadernos Brasileiros de Terapia Ocupacional/Brazilian Journal of Occupational Therapy 2017;25(4):825-37
- [Background] Cohen D, Allen J, Rhydderch M, Aylward M. The return to work discussion: a qualitative study of the line manager conversation about return to work and the development of an educational programme. J Rehabil Med. 2012 Jul;44(8):677-83. doi: 10.2340/16501977-0996. PMID 22729796
- [Background] Scott W, Chilcot J, Guildford B, Daly-Eichenhardt A, McCracken LM. Feasibility randomized-controlled trial of online Acceptance and Commitment Therapy for patients with complex chronic pain in the United Kingdom. Eur J Pain. 2018 Apr 28. doi: 10.1002/ejp.1236. Online ahead of print. PMID 29704880
- [Background] Coutu MF, Legare F, Durand MJ, Stacey D, Labrecque ME, Corbiere M, Bainbridge L. Acceptability and Feasibility of a Shared Decision-Making Model in Work Rehabilitation: A Mixed-Methods Study of Stakeholders' Perspectives. J Occup Rehabil. 2019 Mar;29(1):128-139. doi: 10.1007/s10926-018-9770-1. PMID 29663111
- [Background] Braillard O, Cedraschi C, Jesaimani A, Piguet V. [Chronic noncancer pain and patient education: a place for e-learning?]. Rev Med Suisse. 2015 Jun 24;11(480):1400, 1402-5. French. PMID 26267947
- [Background] Ledel Solem IK, Varsi C, Eide H, Kristjansdottir OB, Borosund E, Schreurs KMG, Waxenberg LB, Weiss KE, Morrison EJ, Haaland-Overby M, Bevan K, Zangi HA, Stubhaug A, Solberg Nes L. A User-Centered Approach to an Evidence-Based Electronic Health Pain Management Intervention for People With Chronic Pain: Design and Development of EPIO. J Med Internet Res. 2020 Jan 21;22(1):e15889. doi: 10.2196/15889. PMID 31961331
- [Background] Kristjansdottir OB, Fors EA, Eide E, Finset A, Stensrud TL, van Dulmen S, Wigers SH, Eide H. A smartphone-based intervention with diaries and therapist feedback to reduce catastrophizing and increase functioning in women with chronic widespread pain. part 2: 11-month follow-up results of a randomized trial. J Med Internet Res. 2013 Mar 28;15(3):e72. doi: 10.2196/jmir.2442. PMID 23538392
- [Background] Thurnheer SE, Gravestock I, Pichierri G, Steurer J, Burgstaller JM. Benefits of Mobile Apps in Pain Management: Systematic Review. JMIR Mhealth Uhealth. 2018 Oct 22;6(10):e11231. doi: 10.2196/11231. PMID 30348633
- [Background] Garg S, Garg D, Turin TC, Chowdhury MF. Web-Based Interventions for Chronic Back Pain: A Systematic Review. J Med Internet Res. 2016 Jul 26;18(7):e139. doi: 10.2196/jmir.4932. PMID 27460413
- [Background] Slattery BW, Haugh S, O'Connor L, Francis K, Dwyer CP, O'Higgins S, Egan J, McGuire BE. An Evaluation of the Effectiveness of the Modalities Used to Deliver Electronic Health Interventions for Chronic Pain: Systematic Review With Network Meta-Analysis. J Med Internet Res. 2019 Jul 17;21(7):e11086. doi: 10.2196/11086. PMID 31317869
- [Background] Ledel Solem IK, Varsi C, Eide H, Kristjansdottir OB, Mirkovic J, Borosund E, Haaland-Overby M, Heldal K, Schreurs KM, Waxenberg LB, Weiss KE, Morrison EJ, Solberg Nes L. Patients' Needs and Requirements for eHealth Pain Management Interventions: Qualitative Study. J Med Internet Res. 2019 Apr 1;21(4):e13205. doi: 10.2196/13205. PMID 30877780
- [Background] Timmers T, Janssen L, Kool RB, Kremer JA. Educating Patients by Providing Timely Information Using Smartphone and Tablet Apps: Systematic Review. J Med Internet Res. 2020 Apr 13;22(4):e17342. doi: 10.2196/17342. PMID 32281936
- [Background] Granja C, Janssen W, Johansen MA. Factors Determining the Success and Failure of eHealth Interventions: Systematic Review of the Literature. J Med Internet Res. 2018 May 1;20(5):e10235. doi: 10.2196/10235. PMID 29716883
- [Background] Devan H, Hale L, Hempel D, Saipe B, Perry MA. What Works and Does Not Work in a Self-Management Intervention for People With Chronic Pain? Qualitative Systematic Review and Meta-Synthesis. Phys Ther. 2018 May 1;98(5):381-397. doi: 10.1093/ptj/pzy029. PMID 29669089
- [Background] Devan H, Farmery D, Peebles L, Grainger R. Evaluation of Self-Management Support Functions in Apps for People With Persistent Pain: Systematic Review. JMIR Mhealth Uhealth. 2019 Feb 12;7(2):e13080. doi: 10.2196/13080. PMID 30747715
- [Background] Ruckenstein M. Visualized and interacted life: personal analytics and engagement with data doubles. Societies. 2014;4:68-84. doi: 10.3390/soc4010068.
- [Background] Mamykina L, Smaldone AM, Bakken SR. Adopting the sensemaking perspective for chronic disease self-management. J Biomed Inform. 2015 Aug;56:406-17. doi: 10.1016/j.jbi.2015.06.006. Epub 2015 Jun 10. PMID 26071681
- [Background] Morton K, Dennison L, May C, Murray E, Little P, McManus RJ, Yardley L. Using digital interventions for self-management of chronic physical health conditions: A meta-ethnography review of published studies. Patient Educ Couns. 2017 Apr;100(4):616-635. doi: 10.1016/j.pec.2016.10.019. Epub 2016 Oct 20. PMID 28029572
- [Background] Machado GC, Pinheiro MB, Lee H, Ahmed OH, Hendrick P, Williams C, Kamper SJ. Smartphone apps for the self-management of low back pain: A systematic review. Best Pract Res Clin Rheumatol. 2016 Dec;30(6):1098-1109. doi: 10.1016/j.berh.2017.04.002. Epub 2017 May 25. PMID 29103552
- [Background] Coe-O'Brien R, Joseph L, Kuisma R, Paungmali A, Sitilertpisan P, Pirunsan U. Outcome measures used in the smartphone applications for the management of low back pain: a systematic scoping review. Health Inf Sci Syst. 2020 Jan 2;8(1):5. doi: 10.1007/s13755-019-0097-x. eCollection 2020 Dec. PMID 31938540
- [Derived] Turesson C, Liedberg G, Vixner L, Lofgren M, Bjork M. Evidence-based digital support during 1 year after an Interdisciplinary Pain Rehabilitation Programme for persons with chronic musculoskeletal pain to facilitate a sustainable return to work: a study protocol for a registry-based multicentre randomised controlled trial. BMJ Open. 2022 Apr 25;12(4):e060452. doi: 10.1136/bmjopen-2021-060452. PMID 35470201